CLINICAL TRIAL: NCT05741983
Title: A Prospective, Double Blind, Single-centre, Randomised Controlled Trial Comparing Arthroscopic Autologous Matrix Induced Chondrogenesis (AMIC®) to Microfracture Alone in the Treatment of Osteochondral and Chondral Lesion in the Ankle (AMARTA)
Brief Title: AMIC vs. MFx in the Ankle
Acronym: AMARTA
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: unsatisfactory patient enrollment
Sponsor: Geistlich Pharma AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 13575-236
Record Dates: First submitted 2023-02-01; First posted 2023-02-23 (Actual); Last update posted 2024-03-18 (Actual); Status verified 2024-03

CONDITIONS: Osteochondral Lesion of Talus; Chondral Defect; Microfracture
Keywords: double-blind Randomised Controlled Trial (RCT); Chondro-Gide®; AMIC®
MeSH Terms: conditions — Fractures, Stress

STUDY DESIGN:
Intervention Model Description: Double blind RCT (Randomized Controlled Trial)
Who Masked: Participant, Outcomes Assessor
Masking Description: Patients will be blinded to the surgical procedure (with or without membrane). The outcome assessor who will complete the AOFAS and TAS will not be the physician who performed the surgery, the examiner is blinded to the treatment group to which the patient was allocated.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AMIC® (Experimental): Bone Marrow Stimulation (Microfracture) with Chondro-Gide®
  Interventions: Procedure: Microfracture (MFx); Device: Chondro-Gide®
- Microfracture (MFx) (Active Comparator): Microfracture alone
  Interventions: Procedure: Microfracture (MFx)

INTERVENTIONS:
Procedure: Microfracture (MFx) — The ankle arthroscopy will be a standard procedure. The lesion will be identified, measured and prepared with curettage and soft tissue shaver. Preparation includes debridement of the unstable cartilage and in case of a chondral defect associated with a bone defect, the subchondral cyst is debrided. After debridement, the defect is classified and the lesion size is measured again.The microfracture will be performed with a microfracture awl. In cases of a chondral defect associated with a bone defect (osteochondral defect) the bone lesion must be treated concomitantly. Portal closure will be with steri-strips. All patients will follow the standard postoperative rehabilitation protocol including post op non-weight bearing and range of motion exercises for 6 weeks.
Device: Chondro-Gide® — After the microfracture is performed and before the concomitant treatment of a bony lesion (if present), the defect size will be templated, and the membrane cut into its correct size. The joint is then drained and the membrane will be applied over the defect and stabilised with Fibrin glue. In cases of a osteochondral defect the bone lesion must be treated concomitantly. Once the bone defect has been treated, the Chondro-Gide® membrane is used to cover the site, and to support new cartilage tissue formation at the joint interface. Fluid will be reintroduced, and the stability of the membrane will be confirmed arthroscopically.
  Arms: AMIC®

SUMMARY:
This clinical investigation is a prospective, double blind, single-centre, randomised controlled trial comparing arthroscopic autologous matrix induced chondrogenesis (AMIC®) to microfracture alone in the treatment of osteochondral and chondral lesion in the ankle to evaluate effectiveness, performance and safety of AMIC® procedure versus microfracture (MFx).

DETAILED DESCRIPTION:
This clinical investigation compares arthroscopic autologous matrix induced chondrogenesis (AMIC®) to microfracture alone in the treatment of osteochondral and chondral lesion in the ankle to evaluate effectiveness, performance and safety of AMIC® procedure versus microfracture (MFx). It is a prospective, double blind, single-centre, randomised controlled trial. The objective of this clinical investigation is to evaluate performance, effectiveness, and safety of AMIC® procedure versus Microfracture (MFx). The effectiveness of the treatment is measured by the difference in the walking/standing- part score taken from the Manchester Oxford Foot Questionnaire (MOX-FQ) from baseline to 12 months. The secondary endpoints concern clinical safety and performance. Patients will be randomized into two groups: Microfracture alone (MFx) or Bone Marrow Stimulation (Microfracture) with Chondro-Gide® (AMIC®). The investigational device will be assessed within its intended use.

ELIGIBILITY:
Inclusion criteria:

* Signed written informed consent
* Diagnosis of symptomatic osteochondral or chondral lesion of the talus, deemed by surgeon amenable to arthroscopic treatment with debridement and microfracture
* Age of 18-65 years
* Subject is willing and able to comply with all study procedures, including visits, diagnostic procedures, the rehabilitation protocol and responding to patient questionnaire follow up

Exclusion criteria:

* Lesions smaller 1 square centimeters and greater than 4 square centimeters based on the MRI
* Malalignment which is not corrected prior to or as part of same surgery
* Established significant hindfoot arthritis
* Patients who are unable to have an MRI scan
* Chronic inflammatory arthritis or infectious arthritis
* History of autoimmune disease or immunodeficiency
* History of connective tissue disease
* Intra-articular steroid use within the 3 months prior to enrolment
* Other intra-articular injections (e.g., hyaluronic acid) within 3 months prior to enrolment
* The patient is currently being treated with radiation, chemotherapy, immunosuppression, or systemic steroid therapy with a dose equivalent to more than 5 mg prednisolone
* Pregnancy or lactation
* Enrolled in another study, involved in the study (as a researcher/investigator/sponsor), or relative of someone directly involved in the clinical investigation
* Active infection of the index ankle
* Has been prescribed medication to treat osteoporosis
* Any disorder or impairment that would interfere with evaluation of outcomes measures, such as neurological, degenerative muscular, psychiatric, or cognitive conditions

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-04-28 (Actual); Primary Completion 2024-02-06 (Actual); Study Completion 2024-02-06 (Actual)

PRIMARY OUTCOMES:
Manchester Oxford Foot Questionnaire (MOX-FQ) walking/standing subscale | difference from baseline to 12 months post-operative
  The effectiveness of the treatment is measured by the difference in the walking/standing- part score taken from the the MOX-FQ from baseline to 12 months. Raw score values for the walking/standing part are between 0-28, where higher score mean a worse outcome. Raw scores are converted to a metric (0-100).

SECONDARY OUTCOMES:
Manchester Oxford Foot Questionnaire (MOX-FQ) total | change at 12, 24 and 60 months from baseline
  The MOX-FQ is a commonly reported scoring system in the literature with proven acceptability, reliability and responsiveness for assessment of patients undergoing various foot and ankle surgeries. The total score consists of 3 subscales: Pain, Walking/ Standing and Social interaction. Raw score values for the total score are between 0-64, where higher score mean a worse outcome. Raw scores are converted to a metric (0-100).
American Orthopaedic Foot and Ankle-Hind foot Score (AOFAS) | change at 12, 24 and 60 months from baseline
  The AOFAS has been used as a tool to measure the functional outcome after foot and ankle surgery and is often regarded as an essential outcome measure for all clinical studies. The score ranges from 0 - 100, where higher scores mean better outcomes.
Foot Functioning Index (FFI) | change at 12, 24 and 60 months from baseline
  The FFI measures a patient's function in terms of pain, disability, and activity restriction to assess the impact of foot pathology. The index is self-administered and consists of 23 items, each scored 0 - 10, divided into three sub-scales. Higher scores mean decreased function.
Tegner activity scale (TAS) | change at 12, 24 and 60 months from pre-symptomatic score
  The TAS determines a patient's activity level by grading their work and sports-based activity on a scale of 0 to 10. It is a one-item score and has proven its psychometric properties in knee surgery patients.
EuroQol-5 Dimensions 5 Level (EQ5D-5L) | change at 12, 24 and 60 months from baseline
  EQ5D-5L has been shown to be responsive in detecting changes in patient health status after foot and ankle surgery. The EQ5D-5L is widely used as a general health status measures for a wide variety of conditions and enables comparisons of health-related quality of life between different conditions. A summary index is derived from the patients answers, by applying a specific formula.
Magnetic resonance Observation of Cartilage Repair Tissue (MOCART) score | change at 24 and 60 months from baseline
  The MOCART score was originally designed for evaluation of the cartilage in the knee, after procedures like microfracturing, and has a broad use to assess AMIC® in talus. The score is based on nine radiologic variables; degree of repair and defect filling, integration to border tissue, surface and structure of repair tissue, subchondral lamina and bone, adhesions and synovitis. The Score ranges from 0 - 100, where higher scores mean a better outcome.
Safety endpoints | through study completion, an average of 5 years
  Safety will be measured by freedom from device and procedure-related serious adverse events (SADEs) and all other Adverse Events (AEs) or Serious Adverse Events (SAEs) occurred.

CONTACTS AND LOCATIONS:
Overall Officials: Despoina Natsiou Schmiady, Dr., Study Director — Geistlich Pharma AG; Torres Paulo, Mr., Principal Investigator — Freeman Hospital, Newcastle upon Tyne Hospitals NHS Foundation Trust
Locations (1):
- Freeman Hospital, Newcastle upon Tyne, United Kingdom